CLINICAL TRIAL: NCT04641468
Title: Clinical Efficacy and Safety of a Prospective, Multicenter Drug Coated Balloon for Left Main Artery Disease in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-02-002-K01
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Coronary Diseases; Left Main Coronary Artery Disease; Bifurcation Lesions
Keywords: DCB; left main trunk; Bifurcation lesions
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mediana 010 or 001 left main bifurcation lesion (Other): DCB alone combined with retracted DES implantation if necessary (d-p-d strategy)
  Interventions: Procedure: DCB

INTERVENTIONS:
Procedure: DCB — OCT technical guidance: if B-type or C-type dissection can be seen, Oct should be used for further evaluation, and des treatment should be conducted if necessary
  Other Names: optical coherence tomography

SUMMARY:
This is a prospective and observational study. Patients with primary mediana 010 or 001 left main bifurcation lesions were treated with drug ball coated balloon from November 2018 to November 2020 in four hospitals in Huaihai area. The clinical characteristics, pathological changes, operation process and perioperative drug treatment data were collected. Clinical follow-up included hospitalization, postoperative telephone or outpatient follow-up. Objective to compare the safety and efficacy of drug-eluting balloon and drug-eluting stent implantation alone in the treatment of primary mediana 010 or 001 left main bifurcation lesions.

DETAILED DESCRIPTION:
At present, the primary left main trunk end bifurcation lesions with mediana classification of 010 or 001 are mainly treated by crossing stent technique or direct precise positioning stent technology. Because of the difficulty of precise stent placement, the displacement of cristae across stent implantation is easy to affect the distal vessels of the side branch or main branch, and the long-term clinical efficacy is not good, so the standardized interventional therapy is still controversial. Recently, a registered study published by regatelli et al. Showed that spanning stent technology seems to be superior to precise positioning stent technology, but the major adverse cardiac event rate in clinical follow-up is high.

Drug coated balloon (DCB) as a new interventional therapy in recent years, has been gradually used in the treatment of primary coronary artery disease in situ. The latest international consensus on the treatment of coronary heart disease with DCB indicates that more and more clinical studies have shown the safety and effectiveness of DCB in the treatment of coronary artery disease (≥ 3.0 mm). However, there are few studies on the interventional therapy of DCB in the primary mediana type 010 or 001 left trunk end bifurcation lesions, especially the combination of "1-2mm" drug-eluting stent (DES) implantation when necessary.

The purpose of this study was to investigate the feasibility and short-term clinical efficacy of DCB combined with DES implantation in the treatment of primary mediana 010 or 001 left main bifurcation lesions, and to explore a new treatment for such lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non pregnant women aged 18-75 years old;
2. There is clear evidence of myocardial ischemia, including typical ECG changes, non ST segment elevation acute coronary syndrome, ST segment elevation acute myocardial infarction, etc;
3. For mediana 010 or 001 confirmed by coronary angiography, the stenosis was more than 70% by visual inspection and less than 30% at the end of left main artery;
4. They can receive DCB treatment;
5. The reference vessel diameter was 2.00 ~ 4.00 mm;
6. To understand the potential risk of operation and have the intention of DCB treatment.

Exclusion Criteria:

1. Hemodynamic instability, unable to tolerate surgery;
2. The left ventricular ejection fraction was less than 35%;
3. Contrast medium allergy or contraindication for secondary prevention of coronary heart disease;
4. Stents were implanted in the left main trunk;
5. Severe renal insufficiency (EGFR ≤ 30 ml / min / 1.73 m2);
6. Severe infection;
7. Life expectancy is less than one year. All patients signed the informed consent of interventional therapy before operation, and this study was approved by hospital ethics committee.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The patients were followed up for 12 months to observe the major adverse cardiac events (MACE) | 12 months after operation
  There were three endpoints: cardiovascular death, myocardial infarction and stroke

SECONDARY OUTCOMES:
Incidence of target lesion revascularization | 12 months after operation
  Target lesion revascularization
All revascularization rates | 12 months after operation
  All revascularization

CONTACTS AND LOCATIONS:
Overall Officials: yaojun zhang, doctor, Principal Investigator — Head of Cardiology Department of Xuzhou Third People's Hospital
Locations (1):
- Xuzhou Third People's Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Result] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Result] Gruchalla KJ, Nawarskas JJ. The paclitaxel-eluting stent in percutaneous coronary intervention: part I: background and clinical comparison to bare metal stents. Cardiol Rev. 2006 Mar-Apr;14(2):88-98. doi: 10.1097/01.crd.0000200895.60631.0b. PMID 16493246
- [Result] Navarese EP, Austin D, Gurbel PA, Andreotti F, Tantry U, James S, Buffon A, Kozinski M, Obonska K, Bliden K, Jeong YH, Kubica J, Kunadian V. Drug-coated balloons in treatment of in-stent restenosis: a meta-analysis of randomised controlled trials. Clin Res Cardiol. 2013 Apr;102(4):279-87. doi: 10.1007/s00392-012-0532-3. Epub 2012 Dec 20. PMID 23262495
- [Result] Bavry AA, Kumbhani DJ, Helton TJ, Borek PP, Mood GR, Bhatt DL. Late thrombosis of drug-eluting stents: a meta-analysis of randomized clinical trials. Am J Med. 2006 Dec;119(12):1056-61. doi: 10.1016/j.amjmed.2006.01.023. PMID 17145250
- [Result] Stettler C, Wandel S, Allemann S, Kastrati A, Morice MC, Schomig A, Pfisterer ME, Stone GW, Leon MB, de Lezo JS, Goy JJ, Park SJ, Sabate M, Suttorp MJ, Kelbaek H, Spaulding C, Menichelli M, Vermeersch P, Dirksen MT, Cervinka P, Petronio AS, Nordmann AJ, Diem P, Meier B, Zwahlen M, Reichenbach S, Trelle S, Windecker S, Juni P. Outcomes associated with drug-eluting and bare-metal stents: a collaborative network meta-analysis. Lancet. 2007 Sep 15;370(9591):937-48. doi: 10.1016/S0140-6736(07)61444-5. PMID 17869634
- [Result] Hassan AK, Bergheanu SC, Stijnen T, van der Hoeven BL, Snoep JD, Plevier JW, Schalij MJ, Wouter Jukema J. Late stent malapposition risk is higher after drug-eluting stent compared with bare-metal stent implantation and associates with late stent thrombosis. Eur Heart J. 2010 May;31(10):1172-80. doi: 10.1093/eurheartj/ehn553. Epub 2009 Jan 21. PMID 19158118
- [Result] Chang M, Park DW. Optimal Duration of Dual Antiplatelet Therapy After Implantation of Drug-Eluting Stents: Shorter or Longer? Cardiol Ther. 2014 Dec;3(1-2):1-12. doi: 10.1007/s40119-014-0030-y. Epub 2014 Nov 1. PMID 25367504
- [Result] De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E, Juni P; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI for stable coronary artery disease. N Engl J Med. 2014 Sep 25;371(13):1208-17. doi: 10.1056/NEJMoa1408758. Epub 2014 Sep 1. PMID 25176289